CLINICAL TRIAL: NCT00296569
Title: A 4-Week, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of MK0686 in Patients With Osteoarthritis of the Knee or Hip
Brief Title: A Study to Assess the Safety and Efficacy of an Investigational Drug (MK-686) in Patients With Osteoarthritis (0686-006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0686-006; MK0686-006; 2006_011
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — methyl 3-chloro-3'-fluoro-4'-(1-(((1-((trifluoroacetyl)amino)cyclopropyl)carbonyl)amino)ethyl)-1,1'-biphenyl-2-carboxylate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0686

SUMMARY:
This study is being conducted to assess the safety and tolerability of MK-0686 and to evaluate its efficacy in the treatment of osteoarthritis of the hip or knee in men and women.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical and radiographic diagnosis of osteoarthritis of the hip or knee,either prior NSAID or Acetaminophen users within the ARA functional class I,II or III and with no clinically significant diseases
* Patients required to demonstrate a flare of the signs and symptoms of OA following withdrawal of NSAID treatment
* Prior acetaminophen users also required to demonstrate greater than a defined minimum level of signs and symptoms of OA
* females must be either post-menopausal or surgically sterilized

Exclusion Criteria:

* No history of concurrent arthritic disease
* No history of neoplastic disease within a specified duration
* No history of disease that causes malabsorption
* Chronic use of certain medications excluded

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Pain relief at the knee and hip over 4 weeks of treatment as assessed by the WOMAC Pain Subscale. | over 4 weeks of treatment

SECONDARY OUTCOMES:
Safety and tolerability over a 4-week treatment period | over a 4-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC